CLINICAL TRIAL: NCT05453890
Title: The Prevalence of Gingival Pigmentation Among a Sample of Adult Egyptian Population: A Cross Sectional Study.
Brief Title: The Prevalence of Gingival Pigmentation Among a Sample of Adult Egyptian Population.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Peter Onsi Doss Hanna, Principal investigator, Cairo University
Other Study IDs: POD 1
Record Dates: First submitted 2022-07-02; First posted 2022-07-12 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Gingival Pigmentation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A sample of adult egyptian population

SUMMARY:
This observational cross-sectional study aims at determining the prevalence of gingival pigmentation among a sample of adult Egyptian patients attending the diagnostic centre at Faculty of Dentistry, Cairo University and identifying its association with other risk factors.

DETAILED DESCRIPTION:
* Dental patients will be recruited in a consecutive manner from the diagnostic center, Faculty of Dentistry, Cairo University.
* Medical history will be taken and patients with certain diseases as Addison's disease, Albright's syndrome, Hereditary hemorrhagic telangiectasia, and HIV-associated melanosis or under certain drugs as ACTH, Antimalarial drugs, and Chemotherapeutic agent-busulfan that induce gingival pigmentation will be excluded from the study.
* Patients who met the inclusion criteria will be subjected to thorough oral examination and a full questionnaire will be filled for each patient. Before filling the questionnaire, the aim of the study will be explained to the patient and the patient's acceptance to participate in the survey will be received.
* During examining patients, any patient found with suspicious gingival pigmentation, whether the degree of pigmentation, texture, size, or any clinical signs of malignancy, will be referred to the Oral Medicine department for a thorough oral and lymph nodes examination, and biopsy taking if needed. Also, any other suspicious oral lesion noticed will be treated the same way, and a close follow-up for the patient will be done to ensure that the he/she has gone through all possible examination protocols to exclude any possibility of malignancy or abnormal condition that needs intervention.
* During oral examination of included patients, those will be found to have gingival pigmentation will be classified according to the gingival pigmentation index.
* Non-respondent patients or patients refusing to participate will be reported with the cause of their refusal.
* The Questionnaire will be filled through a face-to-face personal interview with the patient using simple, short, easily comprehended questions.
* The Questionnaire will include a section for information about age, gender, occupation, place of birth and current residential area.
* Detailed information about smoking type (cigarette, shisha, Vape, IQOS, or others), Smoking Frequency, Smoking duration (no. of years) will be gathered
* The degree of satisfaction or dissatisfaction with gingival pigmentation, and the willingness to do a surgical or laser procedure to change it will be evaluated by VAS score.
* Conventional oral examination will be held on a dental unit using the light of the unit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients whose age is 18 years old and above.
* Patient consulting in the diagnostic centre, Faculty of Dentistry, Cairo University.
* Provide informed consent.

Exclusion Criteria:

* Systemic diseases and syndromes known to be associated with oral melanin pigmentation, such as Addison's disease, Albright's syndrome, Hereditary hemorrhagic telangiectasia, and HIV-associated melanosis (Peeran et al 2014).
* Patients taking certain drugs that predispose to drug-induced melanin pigmentation, such as: ACTH, Antimalarial drugs, and Chemotherapeutic agent-busulfan (Peeran et al 2014).
* Tattoos of the oral mucosa
* Patients having problem in opening their mouth or undergoing inter-maxillary fixation where oral examination will not be possible.
* Patients diagnosed with psychiatric problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A sample of adult Egyptian patients attending the diagnostic centre at Faculty of Dentistry, Cairo University and identifying its association with other risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of gingival pigmentation | Up to 30 weeks
  Gingival Pigmentation Index which classified pigmentation into 4 scores according to the position and extent of the gingival pigments:
  * Score 0: Absence of pigmentation
  * Score 1: Spots of brown to black color or pigments.
  * Score 2: Brown to black patches but not diffuse pigmentation
  * Score 3: Diffuse brown to black pigmentation, marginal, and attached

SECONDARY OUTCOMES:
Age of the participant associated risk factors | Up to 30 weeks
  Age in years
Gender of the participant | Up to 30 weeks
  Male or female
Occupation of the participant | Up to 30 weeks
  Certain occupations may be a possible risk factor
Type of smoking | Up to 30 weeks
  Cigarette, shisha, Vape, IQOS,… etc. certain types may be of variable risk factor
Frequency of smoking | Up to 30 weeks
  Number of Cigarettes/day, In case of other types: daily, weekly, twice weekly, monthly
Duration of smoking | Up to 30 weeks
  In years
Place of birth | Up to 30 weeks
  City of birth
Current area of residence | Up to 30 weeks
  City of residence

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt